CLINICAL TRIAL: NCT02363686
Title: Aspiration in Acute Respiratory Failure Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0184; 5K24HL089223 (NIH); 1R21NR015886-01 (NIH)
Record Dates: First submitted 2015-01-20; First posted 2015-02-16 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEES & Bedside Swallow Evaluation (BSE) (Other): Subjects will receive a Fiberoptic Endoscopic Evaluation of Swallowing (FEES), followed by a speech language pathologist (SLP) performing a bedside swallowing evaluation (BSE).
  Interventions: Procedure: FEES; Procedure: BSE

INTERVENTIONS:
Procedure: FEES — A thin, flexible endoscope designed for assessment of laryngeal structures is passed through the nose to the oropharynx, visualizing the laryngeal structures, and the base of tongue and the pharynx. If needed 4% topical lidocaine and/or oxymetazoline (Afrin) will be administered. Swallowing will then be evaluated directly with six food boluses of 5 ml each. All patients will be allowed to swallow spontaneously without a verbal command to swallow. Video of the examinations will be recorded and presence of dysphagia will be designated independently by 3 different observers (one pulmonary physician and two speech language pathologists (SLPs)). This procedure will take 5-10 minutes. The camera will then be removed.
  Other Names: Fiberoptic Endoscopic Evaluation of Swallowing
Procedure: BSE — Following the FEES, a speech language pathologist (SLP) will perform a noninvasive bedside swallow evaluation (BSE). The SLP will be blinded to the results of the FEES, and the name of the SLP performing the BSE will not be recorded. No other identifying information will be collected regarding the SLP performing the test.
  Other Names: Bedside Swallowing Evaluation

SUMMARY:
The purpose of this study is to learn more about problems with swallowing that could develop in patients who are very sick and need a machine to help them breathe.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about problems with swallowing that could develop in patients who are very sick and need a machine to help them breathe. Patients are asked to be in this study because they had problems breathing on their own and therefore needed the help of a machine called a ventilator. In order for this ventilator to push air into the lungs, patients need a tube placed in the throat called an endotracheal tube. The process of placing this endotracheal tube was called intubation. The tube has now been removed, which is a process called extubation. Sometimes, people who have had endotracheal tubes can have difficulty swallowing food and liquids for a period of time. This disease is called post-extubation dysphagia (PED). PED is a serious condition and may result in food or liquid going from the mouth into the lungs. This could cause further lung problems. Given this risk, doctors sometimes suggest that patients with PED either avoid eating or drinking, or get a feeding tube. Currently, nobody knows how often patients develop PED, why they develop it, or the best method to detect it. Standard care involves clinicians making educated guesses. This study looks to determine if watching the patient swallow, both with and without a small camera, is an accurate method for detecting PED.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in the study if they meet all of the following criteria:

  1. Admission to a University of Colorado Hospital ICU
  2. Mechanical ventilation support through an endotracheal tube for greater than 24 hours

Exclusion Criteria:

* Subjects will be ineligible to participate in the study if they meet any of the following criteria

  1. Age less than 18 years
  2. Contraindication to enteral nutrition administration
  3. Diagnosis of an acute or pre-existing central nervous system disorder (excluding a seizure disorder)
  4. Pre-existing dysphagia
  5. Previous surgery of the head, neck, or esophagus
  6. Previous cancer of the head or neck
  7. The presence of a tracheostomy
  8. The presence of nasal or pharyngeal trauma or bleeding
  9. Clinical team believes one of the protocols would be harmful to an individual patient
  10. Expected survival less than 3 months
  11. Pregnancy
  12. Imprisoned at the time of admission, anytime during the hospitalization, or anytime during the followup period
  13. Inability to give informed consent and proxy unavailable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2012-02; Primary Completion 2018-08-31 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Boston University Medical Center, Boston, Massachusetts

REFERENCES:
- [Background] Ekberg O, Hamdy S, Woisard V, Wuttge-Hannig A, Ortega P. Social and psychological burden of dysphagia: its impact on diagnosis and treatment. Dysphagia. 2002 Spring;17(2):139-46. doi: 10.1007/s00455-001-0113-5. PMID 11956839
- [Background] Marik PE. Aspiration pneumonitis and aspiration pneumonia. N Engl J Med. 2001 Mar 1;344(9):665-71. doi: 10.1056/NEJM200103013440908. No abstract available. PMID 11228282
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Altman KW, Yu GP, Schaefer SD. Consequence of dysphagia in the hospitalized patient: impact on prognosis and hospital resources. Arch Otolaryngol Head Neck Surg. 2010 Aug;136(8):784-9. doi: 10.1001/archoto.2010.129. PMID 20713754
- [Background] Report on the ASHA Speech-Language Pathology Health Care Survey American Speech-Language-Hearing Association. 2011 SLP health care survey summary report: Number and type ofresponses. Available from: http://www.asha.org/uploadedFiles/HC11-Summary-Report.pdf. 2011; 1-49.
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Behrendt CE. Acute respiratory failure in the United States: incidence and 31-day survival. Chest. 2000 Oct;118(4):1100-5. doi: 10.1378/chest.118.4.1100. PMID 11035684
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Background] Macht M, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Postextubation dysphagia is persistent and associated with poor outcomes in survivors of critical illness. Crit Care. 2011;15(5):R231. doi: 10.1186/cc10472. Epub 2011 Sep 29. PMID 21958475
- [Background] Goldsmith T. Evaluation and treatment of swallowing disorders following endotracheal intubation and tracheostomy. Int Anesthesiol Clin. 2000 Summer;38(3):219-42. doi: 10.1097/00004311-200007000-00013. No abstract available. PMID 10984854
- [Background] Suiter DM, Leder SB. Clinical utility of the 3-ounce water swallow test. Dysphagia. 2008 Sep;23(3):244-50. doi: 10.1007/s00455-007-9127-y. Epub 2007 Dec 4. PMID 18058175
- [Background] Hiss SG, Postma GN. Fiberoptic endoscopic evaluation of swallowing. Laryngoscope. 2003 Aug;113(8):1386-93. doi: 10.1097/00005537-200308000-00023. PMID 12897564
- [Background] Lim SH, Lieu PK, Phua SY, Seshadri R, Venketasubramanian N, Lee SH, Choo PW. Accuracy of bedside clinical methods compared with fiberoptic endoscopic examination of swallowing (FEES) in determining the risk of aspiration in acute stroke patients. Dysphagia. 2001 Winter;16(1):1-6. doi: 10.1007/s004550000038. PMID 11213241
- [Background] O'Neil KH, Purdy M, Falk J, Gallo L. The Dysphagia Outcome and Severity Scale. Dysphagia. 1999 Summer;14(3):139-45. doi: 10.1007/PL00009595. PMID 10341109
- [Background] Aviv JE, Kaplan ST, Thomson JE, Spitzer J, Diamond B, Close LG. The safety of flexible endoscopic evaluation of swallowing with sensory testing (FEESST): an analysis of 500 consecutive evaluations. Dysphagia. 2000 Winter;15(1):39-44. doi: 10.1007/s004559910008. PMID 10594257
- [Background] Cohen MA, Setzen M, Perlman PW, Ditkoff M, Mattucci KF, Guss J. The safety of flexible endoscopic evaluation of swallowing with sensory testing in an outpatient otolaryngology setting. Laryngoscope. 2003 Jan;113(1):21-4. doi: 10.1097/00005537-200301000-00004. PMID 12514376
- [Background] Nacci A, Ursino F, La Vela R, Matteucci F, Mallardi V, Fattori B. Fiberoptic endoscopic evaluation of swallowing (FEES): proposal for informed consent. Acta Otorhinolaryngol Ital. 2008 Aug;28(4):206-11. PMID 18939710
- [Background] Langmore SE, Pelletier C, Nelson. Results of FEES survey on safety of endoscopy for swallowing assessment. Presented at Fourth Annual Meeting of the Dysphagia Research Society, McLean, VA, October 28, 1995.
- [Background] Leder SB, Suiter DM, Warner HL, Acton LM, Siegel MD. Safe initiation of oral diets in hospitalized patients based on passing a 3-ounce (90 cc) water swallow challenge protocol. QJM. 2012 Mar;105(3):257-63. doi: 10.1093/qjmed/hcr193. Epub 2011 Oct 17. PMID 22006561
- [Background] Guidelines and procedures for monitoring VAP. 2011. United States Centers for Disease Control and Prevention (CDC) and National Healthcare Safety Network (NHSN). 22 December 2011. http://www.cdc.gov/nhsn/psc_da.html. 2011; 1-12.
- [Background] Garner JS, Jarvis WR, Emori TG, Horan TC, Hughes JM. CDC definitions for nosocomial infections, 1988. Am J Infect Control. 1988 Jun;16(3):128-40. doi: 10.1016/0196-6553(88)90053-3. PMID 2841893
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Hospital-acquired pneumonia in adults: diagnosis, assessment of severity, initial antimicrobial therapy, and preventive strategies. A consensus statement, American Thoracic Society, November 1995. Am J Respir Crit Care Med. 1996 May;153(5):1711-25. doi: 10.1164/ajrccm.153.5.8630626. No abstract available.
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Chen AY, Frankowski R, Bishop-Leone J, Hebert T, Leyk S, Lewin J, Goepfert H. The development and validation of a dysphagia-specific quality-of-life questionnaire for patients with head and neck cancer: the M. D. Anderson dysphagia inventory. Arch Otolaryngol Head Neck Surg. 2001 Jul;127(7):870-6. PMID 11448365
- [Background] Bousquet J, Knani J, Dhivert H, Richard A, Chicoye A, Ware JE Jr, Michel FB. Quality of life in asthma. I. Internal consistency and validity of the SF-36 questionnaire. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):371-5. doi: 10.1164/ajrccm.149.2.8306032.
- [Background] Chrispin PS, Scotton H, Rogers J, Lloyd D, Ridley SA. Short Form 36 in the intensive care unit: assessment of acceptability, reliability and validity of the questionnaire. Anaesthesia. 1997 Jan;52(1):15-23. doi: 10.1111/j.1365-2044.1997.015-az014.x. PMID 9014540
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Derived] Langmore SE, Krisciunas GP, Warner H, White SD, Dvorkin D, Fink D, McNally E, Scheel R, Higgins C, Levitt JE, McKeehan J, Deane S, Siner JM, Vojnik R, Moss M. Correction to: Abnormalities of Aspiration and Swallowing Function in Survivors of Acute Respiratory Failure. Dysphagia. 2021 Oct;36(5):842-853. doi: 10.1007/s00455-020-10226-8. PMID 33635374
- [Derived] Langmore SE, Krisciunas GP, Warner H, White SD, Dvorkin D, Fink D, McNally E, Scheel R, Higgins C, Levitt JE, McKeehan J, Deane S, Siner JM, Vojnik R, Moss M. Abnormalities of Aspiration and Swallowing Function in Survivors of Acute Respiratory Failure. Dysphagia. 2021 Oct;36(5):831-841. doi: 10.1007/s00455-020-10199-8. Epub 2020 Nov 6. PMID 33156398
- [Derived] Krisciunas GP, Langmore SE, Gomez-Taborda S, Fink D, Levitt JE, McKeehan J, McNally E, Scheel R, Rubio AC, Siner JM, Vojnik R, Warner H, White SD, Moss M. The Association Between Endotracheal Tube Size and Aspiration (During Flexible Endoscopic Evaluation of Swallowing) in Acute Respiratory Failure Survivors. Crit Care Med. 2020 Nov;48(11):1604-1611. doi: 10.1097/CCM.0000000000004554. PMID 32804785
- [Derived] Moss M, White SD, Warner H, Dvorkin D, Fink D, Gomez-Taborda S, Higgins C, Krisciunas GP, Levitt JE, McKeehan J, McNally E, Rubio A, Scheel R, Siner JM, Vojnik R, Langmore SE. Development of an Accurate Bedside Swallowing Evaluation Decision Tree Algorithm for Detecting Aspiration in Acute Respiratory Failure Survivors. Chest. 2020 Nov;158(5):1923-1933. doi: 10.1016/j.chest.2020.07.051. Epub 2020 Jul 25. PMID 32721404
- [Derived] Lynch YT, Clark BJ, Macht M, White SD, Taylor H, Wimbish T, Moss M. The accuracy of the bedside swallowing evaluation for detecting aspiration in survivors of acute respiratory failure. J Crit Care. 2017 Jun;39:143-148. doi: 10.1016/j.jcrc.2017.02.013. Epub 2017 Feb 15. PMID 28259057

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 213 patients were included in the final analysis
Period: Overall Study
Arm/Group | FEES & Bedside Swallow Evaluation (BSE)
Started | 248
Completed | 213
Not Completed | 35
Not completed — Withdrawal by Subject | 22
Not completed — incomplete FEES examinations | 13

BASELINE CHARACTERISTICS:
Arm/Group | FEES & Bedside Swallow Evaluation (BSE)
Number analyzed (Participants) | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 212
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 57 [47 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 131
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 54
  White | 117
  More than one race | 0
  Unknown or Not Reported | 42
Region of Enrollment [Number; unit: participants]
  United States | 213

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Aspiration
Description: Aim: To develop a BSE-based non-invasive clinical prediction rule (CPR) that will accurately and efficiently diagnose aspiration in ARF survivors. Aspiration (PAS score of ≥6) on the FEES with any of the five feedings. This outcome measure will report the percentage of participants experiencing silent and non-silent aspiration, as visualized on the FEES. The FEES is a flexible fiberoptic camera that allows the investigators to visualize the patient swallowing each of the 5 different consistencies of food.
Time Frame: from extubation Day 1 through hospital discharge, expected to be within 28 days
Population: Overall, 213 patients were included in the final analysis.
Measure: Number; unit: percentage of participants
Groups:
- FEES & Bedside Swallow Evaluation (BSE): A speech language pathologist (SLP) will perform a bedside swallowing evaluation (BSE).followed by a Fiberoptic Endoscopic Evaluation of Swallowing (FEES). BSE: Before the FEES, a speech language pathologist (SLP) will perform a noninvasive bedside swallow evaluation (BSE). The SLP will be blinded to the results of the FEES, and the name of the SLP performing the BSE will not be recorded. No other identifying information will be collected regarding the SLP performing the test FEES: A thin, flexible endoscope designed for assessment of laryngeal structures is passed through the nose to the oropharynx, visualizing the laryngeal structures, and the base of tongue and the pharynx. If needed 4% topical lidocaine and/or oxymetazoline (Afrin) will be administered. Swallowing will then be evaluated directly with five food boluses of 5 ml each. All patients will be allowed to swallow spontaneously without a verbal command to swallow. Video of the examinations will be recorded and presence of dysphagia will be designated independently by 3 different observers (one pulmonary physician and two speech language pathologists (SLPs)). This procedure will take 5-10 minutes. The camera will then be removed.
  .
Arm/Group | FEES & Bedside Swallow Evaluation (BSE)
Number analyzed (Participants) | 213
percentage of participants
  Overall aspiration | 70
  Non-silent aspiration | 52

ADVERSE EVENTS:
Time Frame: Through study completion, about 28 days
Arm/Group | FEES & Bedside Swallow Evaluation (BSE)
All-Cause Mortality (participants affected / at risk) | 0/248
Serious Adverse Events (participants affected / at risk) | 0/248
Other Adverse Events (participants affected / at risk) | 3/248
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FEES & Bedside Swallow Evaluation (BSE) (N=248)
Vomiting (Gastrointestinal disorders) | 2 (2) — Subject vomited the night of the BSE and FEES
GI bleed (Gastrointestinal disorders) | 1 (1) — subject re-intubated same day after GI bleed
penetration (Gastrointestinal disorders) | 1 (1) — stopped study due to penetration combined with vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02363686/Prot_SAP_000.pdf